CLINICAL TRIAL: NCT05029583
Title: A Cluster Randomized Trial to Determine Diagnostic and Clinical Outcomes From Enhanced SCREENing Strategies for NASH in Type 2 Diabetes (SCREEN NASH T2D)
Brief Title: Clinical Outcomes From Enhanced SCREENing Strategies for NASH in Type 2 Diabetes (SCREEN NASH T2D)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SCREEN NASH T2D
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Nonalcoholic Steatohepatitis; Type 2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The care provider is masked to the primary outcome of the study, but not masked to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine screening group (Experimental): consists of 4 clusters randomized into Group 1 (includes different clinic sites from Group 2)
  Interventions: Other: routine screening
- physician-driven screening group (Active Comparator): consists of 4 clusters randomized into Group 2 (includes different clinic sites from Group 1)
  Interventions: Other: physician-driven screening

INTERVENTIONS:
Other: routine screening — routine screening for advanced NASH
  Arms: routine screening group
Other: physician-driven screening — physician-driven screening for advanced NASH
  Arms: physician-driven screening group

SUMMARY:
The study is stratified cluster randomized trial. The study population will include adults with T2D and presumed NASH.

DETAILED DESCRIPTION:
The study is a multi-centered, stratified cluster randomized controlled, open-labeled two-phase study. Clusters will be independent LMC clinic sites with patients as participants. The use of the stratified cluster randomization design will help prevent the potential for cross-contamination of screening methods.

Study participants who meet eligibility criteria undergo NASH screening. Everything, other than routineness of screening, is maintained the same in both the groups. The screening intervention received is determined by the site of the participant's provider. All participants enrolled will undergo biochemical screening. Regardless of randomization, any participants meeting biochemical cut-offs (FIB-4 index ≥1.3 or NFS >-1.455) will undergo FibroScans. Clinical data and a health-related quality of life assessment will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2D
* Age 18 - 80 years
* BMI >25 kg/m2 or waist circumference ≥102 cm in men and ≥88 cm in women
* Informed consent

Exclusion Criteria:

* Known history of biopsy-proven NAFLD or NASH, hepatitis B, hepatitis C, HIV, liver cirrhosis, hemochromatosis, drug-induced hepatitis, alcohol-related or autoimmune hepatic disease, history of hepatic decompensation, solid organ transplant, or primary liver cancer, based on electronic medical record
* History of alcohol abuse (≥30 g/day or ≥3 drinks/day for males and ≥20 g/day or ≥2 drinks/day for females)
* Unstable patients with T2D (e.g. end stage renal disease on dialysis, late stage cancer, acute cardiovascular event or any hospitalization in the past 3 months). Note - Emergency room visit without hospitalization is not exclusionary
* Pregnancy/lactation
* Presence of implanted electronic medical device (i.e., pacemaker, as FibroScan cannot be performed)
* Language barriers (i.e. inability to read the consent form translated in any of the multiple languages)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-10-05 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of presumed advanced NASH based on biochemical and FibroScan results | 3 months
  Percent of participants identified with presumed advanced NASH. Specific details for calculating the primary outcome of this study are blinded for health care providers, and therefore not disclosed in this description.

SECONDARY OUTCOMES:
Proportion of study participants with presumed high grade fibrosis | 3 months
  Proportion of study participants with presumed any NASH (fibrosis-4 index >2.67 or NAFLD fibrosis score >0.675 AND FibroScan LSM ≥ 8.0 kPa)
Proportion of study participants with presumed any NASH | 3 months
  Proportion of study participants with presumed any NASH (fibrosis-4 index ≥1.3 or NAFLD fibrosis score >-1.455 AND FibroScan diagnosis of any stage fibrosis)
Proportion of study participants with presumed F2/F3 NASH | 3 months
  Proportion of study participants with presumed F2/F3 NASH (fibrosis-4 index ≥1.3 or NAFLD fibrosis score >-1.455 AND FibroScan diagnosis of F2/F3 fibrosis)
Proportion of study participants with a fibrosis-4 index (FIB-4) and/or NAFLD fibrosis score (NFS) above cut-off values | 1 day
  Proportion of study participants with a fibrosis-4 index (FIB-4) and/or NAFLD fibrosis score (NFS) above cut-off values (FIB-4 ≥1.3 or/and NFS >-1.455)
Proportion of study participants with a fibrosis and/or steatosis (stages) | 1 day
  Proportion of study participants with a fibrosis and/or steatosis (stages) based on FibroScan results
Alcohol consumption by study arm - drinks per day | 1 day
  Alcohol consumption measured as self-reported average drinks per day
Alcohol consumption by study arm - drinks per week | 1 day
  Alcohol consumption measured as self-reported average drinks per week
Alcohol consumption by study arm - Alcohol Use Disorders Identification Test (AUDIT) score | 1 day
  Alcohol consumption measured with the Alcohol Use Disorders Identification Test (AUDIT). AUDIT scores range from a minimum score of 0 to a maximum score of 40, with higher scores indicating a worse outcome.
Health-related quality of life by study arm | 1 day
  Health-related quality of life determined by the chronic liver disease questionnaire for non-alcoholic steatohepatitis (CLDQ-NASH) calculated as total CLDQ-NASH score. The CLDQ-NASH instrument includes 36 items grouped into six domains: abdominal symptoms; activity/energy; emotional health; fatigue; systemic symptoms; and worry. The average of the domain scores (min: 1, max: 7) yields the total CLDQ-NASH score. The minimum possible total score is 1 and the maximum possible total score is 7, with a higher total score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Harpreet Bajaj, MD, Principal Investigator — LMC Diabetes & Endocrinology Ltd.
Locations (1):
- LMC Diabetes & Endocrinology Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No